CLINICAL TRIAL: NCT01252368
Title: Human Intestinal Amino Acid Absorption and the Role of a Local (Renin)-Angiotensin System (RAS)
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: EK-1744
Record Dates: First submitted 2010-11-30; First posted 2010-12-03 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Healthy Participants; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- RAS active drugs: ACE inhibitors and sartanes
  Interventions: Biological: hypertension
- healthy participants

INTERVENTIONS:
Biological: hypertension — patients taking daily ACE inhibitors or sartanes
  Groups: RAS active drugs

SUMMARY:
Aim of this trial is to investigate the expression and localisation of different amino acid transporters and their regulatory proteins derived from the regulatory proteins of the local renin angiotensin system (RAS) in the intestine. This is investigated on one hand in patients who do not take any drugs interfering with RAS. On the other hand expression analysis is done in patients taking daily RAS-active drugs, like ACE inhibitors or sartanes.

After obtaining informed consent of patients attending the hospital for clarification of gastrointestinal symptoms by gastroduodenoscopy or colonoscopy, 2 biopsies (in addition to biopsies needed for clinical diagnostics) will be taken from each duodenum, jejunum, ileum and descending colon.

Biopsies are investigated anonymously at the Institute of Physiology of the University of Zurich. The mRNA content of amino acid transporters and regulatory proteins, respectively, in the biopsies is analyzed by quantitative PCR. Transport proteins are in addition analyzed with immunohistochemistry.

Furthermore amino acid concentration in plasma and urine samples are analyzed by HPLC. From plasma and serum samples RAS parameters like renin, aldosterone, ACE and angiotensin(1-7) are measured.

ELIGIBILITY:
Inclusion criteria:

* Men and women aged 18-80 years
* BMI 18-35 kg/m2
* Group 1: patients taking daily RAS-active drugs, like ACE inhibitors or sartanes (treatment indication outside of this study)
* Group 2: no therapy with RAS-active drugs, like ACE inhibitors or sartanes Gastroduodenoscopy and/or colonoscopy with a treatment indication outside of this study
* Informed consent

Exclusion criteria:

* Severe pathologic alterations in the gastrointestinal tract (ulcers, tumors, celiac disease; GERD and gastritis are no exclusion criteria)
* Status after operations of the gastrointestinal tract (except uncomplicated appendectomy or inguinal hernia repair)
* Patients with malignant diseases
* Severe acute or chronic diseases which require treatment (e.g. renal replacement therapy)
* Patients with increased bleeding risk (e.g. oral anticoagulation, coagulopathy)
* Drug or alcohol abuse
* Mental disorders which limits the ability to fulfil all study requirements

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients attending the hospital for clarification of gastrointestinal symptoms by gastroduodenoscopy or colonoscopy
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2009-12; Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Werner Schwizer, Professor MD, Principal Investigator — University Hospital Zurich, Gastroenterology and Hepatology
Locations (1):
- University Hospital Zurich, Gastroenterology and Hepatology, Zurich, Canton of Zurich, Switzerland